## **Informed Consent for Patients**

Title: A Randomized Controlled Trial on the Application of Artificial Intelligence (AI) in Skin Assessment for Pressure Injury Prevention and Staging by Critical Care Nurses

NCT Number: Not Available as yet

Document Date
December 5, 2025

# GENERAL CONSENT FOR PARTICIPATION IN RESEARCH موافقة عامة بالمشاركة في بحث

**Title of Research:** A Randomized Controlled Trial on the Application of Artificial Intelligence (AI) in Skin Assessment for Pressure Injury Prevention and Staging by Critical Care Nurses

عنوان البحث: تجربة سريرية عشوانية مضبوطة حول تطبيق النكاء الاصطناعي في تقييم الجلد للوقاية من تقرحات الفراش وتحديد مراحلها من بواسطة ممرضي وحدات العناية المركزة

#### Part I - Research Participant Information Sheet:

الجزء الأول - معلومات للمشارك في البحث:

You are invited to participate in a Scientific research project

أنت مدعو للمشاركة في بحث علمي

Purpose of the Research: is to examine the effectiveness and impact of Al-assisted skin assessments and Pl staging in critical care settings, by comparing its accuracy, reliability, and nurses' confidence and knowledge with those of traditional assessment methods employed by critical care nurses.

أ. الغرض من البحث: تهدف هذه الدراسة إلى تقييم فعالية وتأثير التقييمات المجلدية المدعومة بالذكاء الاصطناعي وتحديد مراحل تقرحات الفراش في وحدات العناية المركزة، من خلال مقارنة دقتها وموثوقيتها ونقة الممرضين ومعرفتهم بها مع طرق التقييم التقليدية التي يستخدمها ممرضو العناية الم كذة

#### B. Description of the Research:

If you agree to take part in this study, nurses will check your skin for any problems such as redness or breaks in the skin. This skin check is part of your usual nursing care, and it involves looking at areas of skin that are more likely to be affected, such as your back, sacrum (lower back), heels, or other pressure points. Each skin check will take about 10–15 minutes and will be done twice during every nursing shift, and more often if there are changes in your skin condition.

For research purposes, the nurses will be divided into two groups. In the first group, nurses will assess your skin in the standard way, by looking and gently touching the skin. In the second group, nurses will also use a special Artificial Intelligence (AI) device. This involves taking a picture of the area being checked, which will then be analyzed by the AI tool to help with the assessment.

In both groups, a wound care specialist will review the results to make sure the most accurate findings are used to guide your treatment plan.

The pictures taken with the AI device will not include your face or any personal information. They will be uploaded to the cloud, where all images will be deidentified so they cannot be traced back to you. The images taken by the nurse will be on a hospital device and will be stored securely and will not be shared outside the study team.

#### ب. وصف البحث:

إذا وافقت على المشاركة في هذه الدراسة، سيقوم الممرضون بفحص بشرتك للتأكد من عدم وجود أي مشكلات مثل الاحمرار أو تشققات الجلد. يُعتبر هذا الفحص جزءًا من رعايتك التمريضية الروتينية، ويتضمن التركيز على المناطق الأكثر عرضة للتأثر مثل الظهر، ومنطقة العَجْز (أسفل الظهر)، والكعبين، أو أي مناطق اخرى معرضة لتقرحات الفراش. يستغرق كل فحص جلدي حوالي 10–15 دقيقة وسيبجرى مرتين خلال كل نوبة تمريضية، وقد يُكرر بشكل أكثر في حال وجود تغييرات في حالة بشرتك. لأغراض البحث، سيتم تقسيم الممرضين إلى مجموعتين. في المجموعة الأولى، سيقيم الممرضون بشرتك بالطريقة المعتادة، من خلال النظر ولمس الجلد برفق. أما في المجموعة الثانية، فسيستخدم الممرضون جهازًا خاصاً الجلد برفق. أما في المجموعة الثانية، فسيستخدم الممرضون جهازًا خاصاً يعتمد على الذكاء الاصطناعي بتحليل الصورة للمساعدة في يقم فحصمها، ثم يقوم نظام الذكاء الاصطناعي بتحليل الصورة للمساعدة في التقييم.

في كلا المجموعتين، سيقوم اخصاني العناية بالجروح بمراجعة النتائج للتاكد من استخدام ادق النتائج الممكنة لتوجيه خطة علاجك. لن تتضمن الصور الماخوذة بواسطة جهاز الذكاء الاصطناعي وجهك أو أي

لن تتضمن الصور الماخودة بواسطه جهاز الدكاء الاصطناعي وجهك او اي معلومات شخصية تخصك. وسيتم تحميل الصور إلى نظام سحابي بعد إزالة جميع البيانات التي قد تُعرَف بك، بحيث لا يمكن ربطها بك. تُحفظ الصور التي يلتقطها الممرض على جهاز تابع للمستشفى بشكل آمن، ولن تتم مشاركتها خارج فريق الدراسة.

المشاركة في هذه الدراسة لن تؤخر أو تغيّر علاجك المعتاد. ستظل رعايتك دائمًا قائمة على أدق وأفضل التقييمات المتاحة.

This Informed Consent Form (ICF) is approved by the KFSHRC IRB

ICF Version No.: 1.0

悉

IRB # 2251201 Approval Dated:

From: 27 October 2025

To: 31 August 2026

INFORMED CONSENT FOR RESEARCH (Cross out the nonapplicable)\*

إذن ناف للجهالة بالموافقة على بحث (اشطب ما لا ينطبق) \*

Participation in this study will not delay or change your normal treatment. Your care will always be based on the most accurate and appropriate assessment available.

#### C. Potential Benefits:

You may not receive a direct benefit from being in this study, since all patients will continue to get the same routine skin care. However, the information we learn may help nurses in the future. The study will show whether using Artificial Intelligence (AI) can make skin checks more accurate and help prevent skin problems such as redness or breaks from becoming worse. The results may also guide hospitals to improve nurse training and develop better ways to keep patients' skin healthy.

#### D. Potential Risks and Discomforts:

This study does not involve any extra medical procedures beyond your usual skin care. Nurses will check your skin in the same way they normally do, so no additional discomfort is expected. If you are in the group where pictures are taken, you may feel a little uneasy about showing the skin that needs to be photographed, but this will only include areas normally checked for skin problems such as your back, sacrum, or heels.

The photographs will not include your face or any personal details. They will be uploaded to the cloud system, and all images will be de-identified so they cannot be linked back to you. The pictures taken by nurses will be stored safely and will not be shared outside the study team.

#### E. Voluntary Participation:

Participation in this study is voluntary. You will not suffer penalty nor loss of any benefits to which you are entitled for,if you decide not to participate.

Significant new findings developed during the course of the study, which might be expected to affect your willingness to continue to participate in the study, will be provided to you.

A signed copy of consent form will be given to you.

# ج. الفوائد المحتملة:

قد لا تحصل على فائدة مباشرة من مشاركتك في هذه الدراسة، لأن جميع المرضى سيستمرون في الحصول على نفس الرعاية الروتينية للبشرة. ومع ذلك، فإن المعلومات التي سنتعلمها قد تساعد الممرضين في المستقبل. ستوضح الدراسة ما إذا كان استخدام الذكاء الاصطناعي (AI) يمكن أن يجعل فحو صات الجلد أكثر دقة ويساعد في منع المشكلات الجلدية مثل الاحمرار أو التشققات من التفاقم. كما قد تُسهم النتائج في توجيه المستشفيات لتحسين تدريب الممرضين وتطوير طرق أفضل للحفاظ على صحة بشرة المرضى.

## د. المخاطر والانزعاجات المحتملة:

هذه الدراسة لا تتضمن أي إجراءات طبية إضافية تتجاوز رعايتك الروتينية للبشرة, سيقوم المعرضون بفحص بشرتك بالطريقة المعتادة نفسها، لذلك لا للبشرة, سيقوم المعرضون بفحص بشرتك بالطريقة المعتادة نفسها، لذلك لا يُتوقع حدوث أي إز عاج إضافي. إذا كنت ضمن المجموعة التي يتم فيها التقاط الصور، فقد تشعر ببعض عدم الارتياح عند إظهار المنطقة الجلاية المراد تصويرها، ولكن التصوير سيقتصر فقط على المناطق التي يتم فحصها عادةً لمشكلات الجلد مثل الظهر، منطقة العَجْز (أسفل الظهر)، أو الكعبين. لن تتضمن الصور وجهك أو أي تفاصيل شخصية. وسيتم تحميلها على النظام السحابي بعد إز الة جميع البيانات التي قد تُعرّف بك، بحيث لا يمكن ربطها بك. كما سيتم حفظ الصور التي يلتقطها الممرضون بشكل آمن، ولن تتم مشاركتها خارج فريق الدراسة.

#### ه. المشاركة الطوعية:

المشاركة في هذه الدراسة طوعية وإذا قررت عدم المشاركة فإنك لن تتعرض لأية مضايقات أو لفقدان حقك المشروع في المعالجة.

سيتم ابلاغك بأية نتائج جديدة هامة تظهر خلال سير الدراسة والتي قد تؤثر في رغبتك في الاستمرار بالمشاركة في هذه الدراسة .

سيتم تزويدك بنسخة موقعة من هذا الإقرار.

This Informed Consent Form (ICF) is approved by the KFSHRC IRB

ICF Version No.: 1.0

AB

IRB # 2251201 Approval Dated:

From: 27 October 2025

To: 31 August 2026

INFORMED CONSENT FOR RESEARCH

(Cross out the nonapplicable)\*

إذن ناف للجهالة بالموافقة على بحث (اشطب ما لا ينطبق) \*

### F. Alternative to Participation (if applicable):

Withdrawal from or not participating in this research study will not affect your ability to obtain alternative methods of medical care available at King Faisal and Research Centre (General Organization) - Jeddah

#### G. Termination of Participation (where applicable):

Taking part in this study is completely voluntary. You have the right to stop participating at any time, for any reason, and this will not affect the care or treatment you receive at the hospital. If you choose to withdraw, any information or pictures collected up to that point may still be used in the study, but no further information will be taken from you.

#### H. Confidentiality:

Your identity and medical record, as a participant in this research study, will remain confidential with respect to any publications of the results of this study. However, your medical record may be reviewed by the principal investigator/ delegate involved in this research, the Research Ethics Committee, or the agency sponsoring this research in accordance with applicable laws and regulations. All pictures taken of the skin will be done so without no identifying information, and will used for the purpose of the assessments only.

#### I. Compensation/ Treatment:

In the event of injury resulting from participation in this research study, KFSHRC-J will make available to you, including admission, if required, its hospital facilities and professional attention. Financial compensation from KFSHRC-J, however, is not available.

#### J. Cost/s Reimbursements:

There will be no cost to you for taking part in this study. All care and skin checks are part of your normal hospital treatment, and you will not be charged for anything related to the study. You will not receive payment for

و. البدائل عن المشاركة (إن وجد):

إن قرارك بعدم الإشتراك أو بالانسحاب من الدراسة لن يؤثر على تلقيك لخدمات علاجية بديلة متو فرة في مستشفى الملك فيصل التخصصي و مركز الابحاث بجدة (مؤسسة عامة).

# ز. إنهاء المشاركة (عند الضرورة):

المشاركة في هذه الدراسة اختيارية بالكامل. لديك الحق في التوقف عن المشاركة في أي وقت ولأي سبب، وإن يؤثر ذلك على الرعاية أو العلاج الذي تتلقاه في المستشفى. إذا اخترت الانسحاب، فقد تُستخدم المعلومات أو الصور التي جُمعت حتى تلك اللحظة ضمن الدراسة، ولكن لن يتم جمع أي معلومات إضافية منك بعد ذلك.

## ح. السرية:

كمشارك في هذه الدراسة ستكون هويتك ومحتويات ملفك الطبي سرية في جميع المنشورات المتعلقة بنتائج الدراسة. إلا إنه يمكن لكل من الباحث الرئيسي/نائبه،أو لجنة أخلاقيات الأبحاث،أو الجهة الداعمة للدر اسة الاطلاع على ملفك الطبى و ذلك في حدود النظم والقوانين المطبقة بهذا الخصوص. سيتم التقاط جميع الصور للجلد دون أي معلومات تعريفية، وستستخدم حصريًا لأغراض التقييم الطبي فقط.

## ط. التعويضات/ العلاج:

في حالة حدوث أي ضرر لا قدر الله من جراء مشاركتك بهذه الدراسة؛ سيتكفل مستشفى الملك فيصل التخصصي ومركز الأبحاث بجدة بتقديم العناية الطبية اللازمة أو التنويم في المستشفى إن لزم الأمر، ولكنه لا يوجد أي تعويضات مالية.

ي التكاليف/ التعويض المالي: لن تتحمل أي تكاليف مقابل مشاركتك في هذه الدراسة. فجميع الرعاية وَفَحُوصِاتَ الْجَلْدُ هِي جَزَّءَ مِن عَلَّاجِكُ الرَّوْتِينِي فِي المُسْتَشْفَى، وَلَن يَتَم فرض أي رسوم عليك تتعلق بالدراسة. كما أنك لن تتلقى أي مقابل مالي مقَّابل المشَّاركة، إلا أن مشاركتك قد تُسهم في تحسين رعاية المرضى في

This Informed Consent Form (ICF) is approved by the KFSHRC IRB

IRB # 2251201 Approval Dated ICF Version No.: 1.0

From: 27 October 2025

To: 31 August 2026

إذن ناف للجهالة بالموافقة على بحث (اشطب ما لا ينطبق) \*

participation, but your involvement may help improve patient care in the future.

#### K. Contact Person(s):

For any specific questions regarding this study or in the event of a research-related injury, please contact the pricipal investigator/delegate, , **Dr Jennifer de Beer** 

phone No. 012667-7777 Ext. 66403

For general questions concerning research at KFSHRC-Jeddah, you may call the research coordinator telephone # 012667-7777

Ext...63537. or the Research Ethics Committee telephone#+966114424528.

## ك. الأشخاص الذين يمكن الاتصال بهم:

في حالة وجود أسئلة محدّدة تتعلّق بهذا البحث ، أو في حالة حدوث أي إصابات تتصل بالدراسة ناتجة عن المشاركة بالدراسة ، نرجو الاتصال على الباحث الرئيسي/نانبه. دكتورة / جيئيفر دي بير هاتف رقم ١٢٦٦٧٧٧٧٠ .

## ل. إقرار الباحث الرنيس لنانبه:

# اقر انا دكتورة / جينيفر دي بير

بانني قد شرحت (للمتطوع/ أو ولي أمره الشرعي)\* المذكور أعلاه بصورة كاملة طبيعة وأهداف مشروع البحث المذكور والمتضمن عدم وجود فائدة مباشرة على المشارك\* والي أي مدى (إن وجد) هي دراسة تجريبية, كما قد شرحت المضاعفات المحتمل حدوثها من جراء هذه الدراسة سواء كانت لأسباب معروفة أو غير معروفة والعواقب والمخاطر المترتبة (إن وجدت) إذا قرر المتطوع إنهاء مشاركته بالدراسة.

كما إنه من المفهوم لدي بأنه قد فهم طبيعة الدراسة والغرض منها والمخاطر الناتجة عنها وذلك قبل توقيعه على الموافقة بالمشاركة ، ولقد قمت بتوضيح استعدادي للإجابة على أي أسئلة متصلة بهذه الدراسة ، وقمت فعلاً بالإجابة الشافية على جميع أسئلته المتعلقة بالدراسة.

## L. I, the principal investigator/delegate

I Dr / Jennifer de Beer have fully explained to the above (volunteer/ guardian)\* the nature and purpose of the above-mentioned research program (including the fact that the studies will not result in any direct therapeutic benefit and the extent, if any, to which the studies are experimental), the possible complications which may arise from both known and unknown causes as a result thereof and the consequences and risks, if any, if the volunteer decides to discontinue participation.

It is my understanding that he/she understands the nature, purposes, and risks of these studies before he signs this informed consent. I have also offered to answer any questions relating to these studies and have fully and completely answered all such questions.

This Informed Consent Form (ICF) is approved by the KFSHRC IRB

ICF Version No.: 1.0

悉

IRB # 2251201 Approval Dated:

From: 27 October 2025

To: 31 August 2026

### PART II: Authorization of Voluntary participant:

# الجزء الثاني: تفويض من المشارك بالدراسة:

M. I, the the participate acknowledge that I have read (or it had been explained to me in a clear language) the attached Research Participant Information Form and **Dr/ Jennifer de Beer** 

has explained to me the nature and purpose of this study in this form, as well as any reasonably expected benefits, possible alternative methods of treatment, the attendant discomforts and risks reasonably expected, and the possibility that complications from both known and unknown causes may arise as a result thereof. I have had the opportunity to ask any questions I had regarding this study and all those questions were answered to my satisfaction. I also agree that blood, body fluids/tissues, and fetus tissues may be sampled for research analyses and related purposes as detailed in the first section of this document.

I acknowledge I do not have any preexisting medical or emotional problem which would make it unwise for me to participate in these studies.

Based on the above mentioned information I voluntarily accept participation in this research study and I understand that I am free to withdraw this consent and discontinue my participation in this study at any time. The consequences and risks, if any, which might be involved if I decided to discontinue my participation have been explained to me. I understand that such withdrawal will not affect my ability to receive any medical care to which I might be otherwise entitled.

م. أقر أنا المشارك بأنني قد قرأت (أو قد شُرحت لي بلغة واضحة) جميع المعلومات الموجودة في نموذج الإقرار بالموافقة على المشاركة بالأبحاث وإن دكتورة / جيئيفر دي بير قد أوضح لي ماهية الدراسة في هذا النموذج, والغرض منها, والفوائد المرجوة منها, والطرق العلاجية البديلة لها, والمخاطر أوالانز عاجات المتوقع حدوثها, وكذلك احتمال حدوث مضاعفات لأسباب معروفة أو غير معروفة نتيجة لذلك. كما أنه قد أتيحت لي الفرصة الكافية لطرح أي سؤال يتعلق بالدراسة وتلقيت الإجابات الكافية. كما أوافق على أنه قد تؤخذ عينات من الدم, سوائل أو أنسجة الجسم, أو أنسجة من الجنين وذلك لأغراض تحليلية ومتعلقة بالبحث كما هو موضح في القسم الاول من هذا المستند.

كما أقر بانني لا أعاني من أي مشاكل طبية أو نفسية معروفة لدي بحيث قد يكون من غير الحكمة أن أشارك بهذه الدراسة.

بناء على ما سبق وبمحض إرادتي فإني أتطوع بالمشاركة في هذه الدراسة, وأفهم أن لي مطلق الحرية بسحب موافقتي وقطع مشاركتي بالدراسة في أي وقت. هذا وقد شرحت لي جميع العواقب والمخاطر المترتبة (إن وجدت) عن انسحابي من الدراسة. كما أفهم بأن انسحابي من هذه الدراسة لن يؤثر في حقي في تلقّي العناية الطبية اللازمة التي أستحقها في الأحوال العادية.

This Informed Consent Form (ICF) is approved by the KFSHRC IRB

ICF Version No.: 1.0

悉

IRB # 2251201 Approval Dated:

From: 27 October 2025

To: 31 August 2026

| Dationt's | Identification | lade l |
|-----------|----------------|--------|

| Title of Research: A Randomized Controlled Trial on the Application of Artificial Intelligence (AI) in Skin Assessment for Pressure Injury Prevention and Staging by Critical Care Nurses | عنوان البحث: |
|---|---|
| Name of Participant: | اسم المشارك: |
| Name of individual signing the consent form: | اسم الموقع على هذا الإقرار: |
| Gaurdian's Relation*: | صفة ولي الأمر *: |
| Signature: | التوقيع: |
| Date: | التاريخ: |
| I confirm that I have accurately (translated and/ or read)* the information to the subject: | أقر بانني قد (قرأت / أو ترجمت) * للمشارك هذه المعلومات بدقة اسم الشاهد : |
| Witness Name: | اسم الساهد : |
| Signature/(National I.D./Iqama/Hospital I.D. No.): | التوقيع/ (رقم الهوية/ الإقامة/ الرقم الوظيفي): |
| Date / Time: | التاريخ/ الوقت: |
| Signature of Principal Investigator/ Delegate | توقيع الباحث الرنيسي/نانبه |
| Name: Dr Jennifer de Beer | الاسم: |
| I.D. No.: 69129 | الرقم الوظيفي: |
| Title:Nursing Research Senior Specialist | الوظيفة: |
| Signature: | التوقيع: |
| Date: | التاريخ: |

This Informed Consent Form (ICF) is approved by the KFSHRC IRB

ICF Version No.: 1.0

悉

IRB # 2251201 Approval Dated:

From: 27 October 2025

To: 31 August 2026